CLINICAL TRIAL: NCT02977429
Title: Clinical Study of Central Venous-to-Arterial Carbon Dioxide Difference(Pcv-aCO2) in the Evaluation of Fluid Therapy for Postoperative Patients With Abdominal Cancer
Brief Title: Evaluation of Pcv-aCO2 in the Fluid Treatment of Abdominal Tumor Patients After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bc2016032
Record Dates: First submitted 2016-10-09; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Abdominal Tumor; Abdominal Infection
Keywords: Tumor; Abdominal infection; Hemodynamics; Pcv-aCO2; Early Goal-directed Therapy (EGDT)
MeSH Terms: conditions — Abdominal Neoplasms; Intraabdominal Infections; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard group (Active Comparator): The patients with ScvO2 ≥ 70% will receive the conventional fluid therapy.than collect the data of ScvO2 and Pcv-aCO2:
  ScvO2≥70%，and furthermore, Pcv-aCO2 is divided into "≤6mmHg" and ">6mmHg"
  Interventions: Other: conventional fluid therapy
- control group (Sham Comparator): The patients with ScvO2 <70% will receive the standardized fluid therapy for 6 hours.than collect the data of ScvO2 and Pcv-aCO2:
  ScvO2<70%，and furthermore, Pcv-aCO2 is divided into "≤6mmHg" and ">6mmHg"
  Interventions: Other: standardized fluid therapy

INTERVENTIONS:
Other: standardized fluid therapy — The patients with ScvO2 <70% will receive the standardized fluid therapy for 6 hours.
  Other Names: Therapeutic effect of fluid resuscitation
  Arms: control group
Other: conventional fluid therapy — The patients with ScvO2 ≥ 70% will receive the conventional fluid therapy.
  Arms: standard group

SUMMARY:
This research will confirm that Pcv-aCO2 is suitable for the guidance of early fluid therapy and the evaluation of the prognosis of patients with abnormal hemodynamics after abdominal tumor surgery, and is expected to be a new monitoring index to improve the therapeutic effect of these patients.

DETAILED DESCRIPTION:
1. Confirmed that Pcv-aCO2 is suitable for the guidance of early fluid therapy and the evaluation of the prognosis of patients with abnormal hemodynamics after abdominal tumor surgery, and is expected to be a new monitoring index to improve the therapeutic efficacy of this kind of patients.
2. Pcv-aCO2 effectively reflected the improvement of tissue and organ microcirculation disorder through the individual goal target treatment to guide the fluid resuscitation in the hemodynamic instability patients.
3. Research of the correlation between Pcv-aCO2 and the organ function in patients with abnormal hemodynamics after operation.

ELIGIBILITY:
Inclusion Criteria:

1. Acute physiology and chronic health score system II (APACHE II) score ≥10；
2. Hemodynamic abnormalities post-operation (a. systolic blood pressure<90mmHg, or descent by basic blood pressure for more than 40mmHg. b. pulse pressure <20mmHg, c. urine volume <0.5ml/Kg/hr, d. heart rate >100 / min, e.Central Venous Pressure(CVP) <5mmHg, f. blood lactic acid >2.7mmol/L, meet any one above).
3. Age ≥ 18 years, which is expected to stay in ICU for 5 days or longer;
4. Patients themselves or their authorized clients agree to participate in clinical trials and signed informed consent.

Exclusion Criteria:

1. age <18 years;
2. without improvement in respiratory system disease or chronic obstructive pulmonary disease with Forced expiratory volume in one second (FEV1) <50%;
3. lobectomy and pneumonectomy;
4. death within 24 after treatment;
5. patients with severe organ dysfunction;
6. pregnant or lactating women;
7. the patients did not sign informed consent;
8. any factors that may be expected to increase the risk of patients or other factors that may interfere with the results of clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-01 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
The change of Pcv-aCO2 | fluid resuscitation for 6 hours, 12 hours and 24 hours
  The change of Pcv-aCO2 (mmHg) after fluid resuscitation for 6 hours, 12 hours and 24 hours respectively.

SECONDARY OUTCOMES:
The treatment success rate in different groups | Twenty-eighth days after admission
  Collect the index of treatment success rate(%) of patients in different groups.
The 28 day mortality in different groups | Twenty-eighth days after admission
  Collect the index of 28 day mortality(%) of patients in different groups.
The hospitalization course in different groups | Twenty-eighth days after admission
  Collect the index of hospitalization course(days) of patients in different groups.

OTHER OUTCOMES:
The change of Central Venous Oxygen Saturation (ScvO2) | fluid resuscitation for 6 hours, 12 hours and 24 hours
  The change of Central venous oxygen saturation (ScvO2, %)after fluid resuscitation for 6 hours, 12 hours and 24 hours respectively.
The change of hemoglobin (Hb) | fluid resuscitation for 6 hours, 12 hours and 24 hours
  The change of hemoglobin (Hb, g/L) after fluid resuscitation for 6 hours, 12 hours and 24 hours respectively.
The change of blood lactic acid (Lac) | fluid resuscitation for 6 hours, 12 hours and 24 hours
  The change of blood lactic acid (Lac, mmol/L) after fluid resuscitation for 6 hours, 12 hours and 24 hours respectively.
The change of Cardiac Index (CI) | fluid resuscitation for 6 hours, 12 hours and 24 hours
  The change of Cardiac Index (CI, L/(min•m^2)) after fluid resuscitation for 6 hours, 12 hours and 24 hours respectively.
The Oxygen Supply status (DO2) in different groups | fluid resuscitation for 6 hours, 12 hours and 24 hours
  Collect the index of oxygen supply (DO2, ml/(min•m^2)) after fluid resuscitation for 6 hours, 12 hours and 24 hours respectively.
The Oxygen Consumption (VO2) in different groups | fluid resuscitation for 6 hours, 12 hours and 24 hours
  Collect the index of oxygen consumption (VO2, ml/(min•m^2)) after fluid resuscitation for 6 hours, 12 hours and 24 hours respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Wanhua Wang, director, Study Director — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Futier E, Robin E, Jabaudon M, Guerin R, Petit A, Bazin JE, Constantin JM, Vallet B. Central venous O(2) saturation and venous-to-arterial CO(2) difference as complementary tools for goal-directed therapy during high-risk surgery. Crit Care. 2010;14(5):R193. doi: 10.1186/cc9310. Epub 2010 Oct 29. PMID 21034476
- [Background] Jones AE, Shapiro NI, Trzeciak S, Arnold RC, Claremont HA, Kline JA; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Lactate clearance vs central venous oxygen saturation as goals of early sepsis therapy: a randomized clinical trial. JAMA. 2010 Feb 24;303(8):739-46. doi: 10.1001/jama.2010.158. PMID 20179283
- [Background] Pope JV, Jones AE, Gaieski DF, Arnold RC, Trzeciak S, Shapiro NI; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Multicenter study of central venous oxygen saturation (ScvO(2)) as a predictor of mortality in patients with sepsis. Ann Emerg Med. 2010 Jan;55(1):40-46.e1. doi: 10.1016/j.annemergmed.2009.08.014. Epub 2009 Oct 25. PMID 19854541
- [Background] Harilall Y, Adam JK, Biccard BM, Reddi A. Correlation between cerebral tissue and central venous oxygen saturation during off-pump coronary bypass graft surgery. Perfusion. 2011 Mar;26(2):83-90. doi: 10.1177/0267659110387846. Epub 2010 Nov 15. PMID 21078769